CLINICAL TRIAL: NCT05901376
Title: MicroRNAs From Blood Samples as Biomarkers for Gastric Cancer Detection: a Diagnostic Study
Brief Title: MicroRNAs From Blood Samples as Biomarkers for Gastric Cancer Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Associate Professor, King Chulalongkorn Memorial Hospital
Other Study IDs: RP023
Record Dates: First submitted 2023-03-29; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer; MicroRNAs
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 cc of blood will be obtained from each subject then the plasma portion will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric Cancer
  Interventions: Diagnostic Test: MicroRNA
- Control
  Interventions: Diagnostic Test: MicroRNA

INTERVENTIONS:
Diagnostic Test: MicroRNA — MiR-20a, MiR-21, MiR-106b, MiR-199a, MiR-223

SUMMARY:
The goal of this observational study is to compare specific microRNA levels from the plasma of gastric cancer patients and healthy volunteers to see if there is an upregulated expression in gastric cancer patients.

The main question it aims to answer is:

- Can microRNAs be effectively used as diagnostic biomarkers for gastric cancer?

Participants will be asked for their consent to obtain 5 cc of blood.

ELIGIBILITY:
Inclusion Criteria for Gastric Cancer group:

* Recently diagnosed gastric cancer
* Never received any treatment for gastric cancer

Inclusion Criteria for Control group:

* Age 50 or above
* Underwent elective upper gastrointestinal endoscopy and negative for gastric cancer
* No prior history of gastric dysplasia or cancer

Exclusion Criteria:

* Patients who cannot give informed consent
* Pregnancy
* Lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from King Chulalongkorn Memorial Hospital
  Inclusion Criteria for Gastric Cancer group:
  * Recently diagnosed gastric cancer
  * Never received any treatment for gastric cancer
  Inclusion Criteria for Control group:
  * Age 50 or above
  * Underwent elective upper gastrointestinal endoscopy and negative for gastric cancer
  * No prior history of gastric dysplasia or cancer
  Exclusion Criteria:
  * Patients who cannot give informed consent
  * Pregnancy
  * Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The different of MiR-20a level between gastric cancer and control group | Day 1
  The different of MiR-20a level between gastric cancer and control group
The different of MiR-21 level between gastric cancer and control group | Day 1
  The different of MiR-21 level between gastric cancer and control group
The different of MiR-106b level between gastric cancer and control group | Day 1
  The different of MiR-106b level between gastric cancer and control group
The different of MiR-199a level between gastric cancer and control group | Day 1
  The different of MiR-199a level between gastric cancer and control group
The different of MiR-223 level between gastric cancer and control group | Day 1
  The different of MiR-223 level between gastric cancer and control group

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Not Required For This Country, Thailand

IPD SHARING:
Plan to Share IPD: No